## COVER PAGE STATISTICAL ANALYSIS PLAN

Title: The College, Alcohol and Peers Study (CAPS)

NCT number: NCT03890484

**Document Date:** 12/11/23

## Statistical Analysis Plan

Descriptive statistics were summarized by means and standard deviations of all variables by condition. Regression analyses were initially proposed to examine the interaction between BSM, group condition (close friends vs new peers), and their interaction to predict number of drinks consumed during ad-lib and changes in BART scores from baseline to pre-alcohol assessments. Due to the fact that study procedures were conducted in groups, our local IRB determined our study increased risk for Covid-19 transmission, we were unable to recruit for 1.5 years during the COVID-19 pandemic of the proposed 2 years of data collection. Thus, the obtained sample size (N=13) was severely limited compared to the proposed sample (N = 100) and based on power analyses, our current sample is not sufficient to address significance of findings. **Thus, no statistical tests were completed and only descriptive results are provided.**